CLINICAL TRIAL: NCT06834841
Title: A Comparative Study Between Dexmedetomidine and Fentanyl As Adjuvants to Hyperbaric Bupivacaine for the Prevention of Post-spinal Shivering in Hip Arthroplasty Surgeries
Brief Title: Dexmedetomidine and Fentanyl As Adjuvants to Hyperbaric Bupivacaine for the Prevention of Post-spinal Shivering in Hip Arthroplasty Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MS147/2024
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-02

CONDITIONS: Post Spinal Shivering
MeSH Terms: interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group D (Active Comparator): For group D, the preservative-free dexmedetomidine 100 μg/ml will be loaded into a 100-unit insulin syringe (1 μg/unit) and 5 units will be added to 4 ml (20 mg) of 0.5% hyperbaric bupivacaine
  Interventions: Drug: Dexmedetomidine
- Group F (Active Comparator): For group F, fentanyl 25 mcg will be given intrathecally added to 4 ml (20 mg) of 0.5% hyperbaric bupivacaine.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — the preservative-free dexmedetomidine 100 μg/ml will be loaded into a 100-unit insulin syringe (1 μg/unit) and 5 units will be added to 4 ml (20 mg) of 0.5% hyperbaric bupivacaine
  Other Names: Precedex
  Arms: Group D
Drug: Fentanyl — Fentanyl (Fentanyl Hameln® 0.1mg/2ml) 25 mcg will be given intrathecally added to 4 ml (20 mg) of 0.5% hyperbaric bupivacaine
  Arms: Group F

SUMMARY:
The aim of this study is to compare the efficacy of intrathecal dexmedetomidine versus intrathecal fentanyl when added to hyperbaric bupivacaine in the prevention of post-spinal shivering in patients undergoing hip arthroplasty surgeries and to observe their effects as regards to sedation and intensity of the block.

DETAILED DESCRIPTION:
Preoperative settings:

All patients fulfilling the inclusion criteria who are undergoing hip arthroplasty surgeries and receiving spinal anaesthesia will be randomised into 2 equal groups, namely group D (Dexmedetomidine group) and group F (Fentanyl group).

Routine pre-operative assessment will be done for all patients including routine history taking, clinical examination, and laboratory investigations (complete blood picture, kidney function tests, liver function tests, prothrombin time, partial thromboplastin time).

An informed written consent will be taken from every patient just before the surgery.

Intraoperative and postoperative settings:

On arrival to the operating room, baseline parameters such as ECG, mean arterial blood pressure, heart rate, and oxygen saturation will be recorded. All the patients will be preloaded with 10 ml/kg of Ringer's solution through peripheral intravenous cannula and monitored with five leads electrocardiography, pulse oximetry, and non-invasive blood pressure (NIBP) (which records systolic, diastolic, and mean blood pressure every 5 min intraoperatively and every 15 min in the recovery room, heart rate was recorded in the same intervals).

Under complete aseptic technique, local anaesthetic in the form of 3 ml of lidocaine 2% will be given at the site of spinal injection. Subarachnoid block will be administered in the sitting position midline approach with 25 gauge (Quincke needle) at L3-L4/L4-L5 space.

For group D, the preservative-free dexmedetomidine 100 μg/ml will be loaded into a 100-unit insulin syringe (1 μg/unit) and 5 units will be added to 4 ml (20 mg) of 0.5% hyperbaric bupivacaine.

For group F, fentanyl 25 mcg will be given intrathecally added to 4 ml (20 mg) of 0.5% hyperbaric bupivacaine.

Patients will be immediately placed in the supine position after completing the spinal block.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, ASA II or ASA III patients scheduled for hip arthroplasty surgeries under spinal anaesthesia.

Age > 20 years.

Exclusion Criteria:

* Patient refusal

  * Patients with known neurologic and psychiatric illness.
  * Contraindications for spinal anaesthesia as bleeding or coagulation test abnormalities, local skin infection at spinal lumbar region, raised intracranial pressure and hypovolemia.
  * Height <150 cm.
  * Systemic disorders like hematological, respiratory, cardiac, renal or hepatic insufficiency.
  * Allergy to any of the drugs used in the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
Post spinal shivering | From injection to 3 hours postoperative
  Post spinal anaesthesia shivering will be graded by a blinded observer during the intraoperative and postoperative period using the scale validated by Crossley and Mahajan, 1994 and Tsai and Chu, 2001:
  0 = no shivering,
  1. = piloerection or peripheral vasoconstriction but no visible shivering,
  2. = muscular activity in only one muscle group,
  3. = muscular activity in more than one muscle group but not generalized shivering,
  4. = shivering involving the whole body. Grades 3, and 4 shivering for at least 3 min will be considered positive, and maximum shivering will be considered if generalized shivering interfering with ECG monitoring. Positive shivering or lower grade shivering will be treated with an IV bolus of pethidine (0.5 mg/kg)

SECONDARY OUTCOMES:
Sedation | From injection to 3 hours postoperative
  Patients will be assessed for sedation using a 4-point sedation score as following:
  0 = Alert or drowsy but easily aroused to an alert state by verbal commands alone.
  1. = sleepy and arousable by verbal commands.
  2. = sleepy and not arousable by verbal stimuli but arousable to a drowsy state by tactile stimuli.
  3. = sleepy and not arousable to a drowsy state by tactile stimuli but can be aroused by painful stimuli
Intensity of the block | From injection to 3 hours postoperative
  Peak sensory level and time to reach this level, time to the first two segment regression, and time to first analgesic rescue will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared once the study is completed